CLINICAL TRIAL: NCT00001964
Title: Treatment of Severe Aplastic Anemia With Combined Immunosuppression: Antithymocyte Globulin (ATG) and Cyclosporine A (CSA), and Mycophenolate Mofetil (MMF)
Brief Title: Combination Therapy of Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000032; 00-H-0032
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Severe Aplastic Anemia
Keywords: Hematopoiesis; Bone Marrow Failure; Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders | interventions — Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- single arm (Experimental): ATG 40 mg/kg/d for 4 d; CsA 2 weeks after at 12 mg/kg/d for 6 months. MMF starting on first day of ATG at 600 mg/m2 twice daily for 18 months
  Interventions: Drug: Cyclosporine A; Drug: ATG; Drug: MMF
- single arm 2 (Experimental): ATG at 40 mg/kg/day for 4 days; MMF at 600 mg/m2 twice daily for 18 months and CsA at 12 mg/kg/day for 6 months starting 2 weeks after ATG and MMF
  Interventions: Drug: Cyclosporine A; Drug: ATG; Drug: MMF

INTERVENTIONS:
Drug: Cyclosporine A — Cyclosporine A
Drug: ATG — ATG
Drug: MMF — MMF

SUMMARY:
This study will test the safety and effectiveness of a combination of three drugs in treating severe aplastic anemia and preventing its recurrence. Two drugs used in this trial ATG and cyclosporine are standard combination therapy for aplastic anemia. This study will try to improve this therapy in three ways: 1) by altering the drug regimen to allow the drugs to work better; 2) by reducing the risk of kidney damage; and 3) by adding a third drug mycophenolate mofetil to try to prevent disease relapse.

Patients with severe aplastic anemia who do not have a suitable bone marrow donor or who decline bone marrow transplantation may participate in this study. Patients will have a skin test for ATG allergy, chest X-ray, blood test, and bone marrow aspiration before treatment begins. ATG will then be started, infused through a vein continuously for 4 days. Ten days after ATG is stopped, cyclosporine treatment will begin, taken twice a day by mouth in either liquid or capsule form and will continue for 6 months. Also, in the first 2 weeks of treatment, patients will be given a full dose of corticosteroid (prednisone) to prevent serum sickness that could develop as a side effect of ATG therapy. The dosage will be decreased after that. Mycophenolate will be started at the same time as ATG, in two daily doses by mouth, and will continue for 18 months.

Patients will be hospitalized at the beginning of the study. During this time, blood will be drawn at 3-week intervals and a bone marrow examination will be repeated 3 months after treatment has begun. Additional tests, including X-rays may be required. After hospital discharge, patients will be followed on an outpatient basis at 3-month intervals. The patients own physician will perform blood tests weekly and kidney and liver function tests every 2 weeks during cyclosporine therapy. Transfusions may be required initially.

DETAILED DESCRIPTION:
Severe acquired aplastic anemia (SAA) has a poor prognosis if untreated. Bone marrow transplantation is available to only a minority of patients due to lack of a matched sibling donor, advanced age of the patient, or cost. Clinical studies at NIH and elsewhere have demonstrated excellent response rates and improved survival with immunosuppressive treatments. Laboratory data implicate underlying cytotoxic T-lymphocyte-mediated suppression of hematopoiesis as the likely proximal cause of disease in most patients. In earlier clinical protocols we treated SAA with cyclosporine A (CSA) (86-H-0007), antithymocyte globulin (ATG) (87-H-0124), and combined ATG and CSA (90-H-0146). While intensive immunosuppression is most effective, relapse is common and some patients also develop second hematologic complications like myelodysplasia. In this protocol, we modify our regimen by delaying the introduction of cyclosporine to promote ATG tolerizing effects and adding mycophenolate mofetil (MMF), a new agent that, like ATG may be relatively specific for activated lymphocytes, in an effort to reduce the high relapse rate.

ELIGIBILITY:
* INCLUSION CRITERIA:

Only patients with SAA will be admitted, defined as:

Bone marrow cellularity less than 30%.

At least two of the following blood count findings: absolute granulocyte count less than 500/mm(3); platelet count less than 20,000/mm(3); reticulocyte count less than 60,000/mm(3).

Age greater than or equal to 1 years.

Weight greater than 12 kg.

EXCLUSION CRITERIA:

Serum creatinine greater than 2 mg/dl or estimated creatinine clearance less than 40 ml/min.

Underlying carcinoma, recent history of radiation or chemotherapy.

Current pregnancy or unwillingness to be treated with oral contraceptives.

Inability to comprehend the investigational nature of the study.

Moribund status or concurrent hepatic, renal, cardiac, neurologic, or metabolic disease of such severity that death within 7 to 10 days is likely.

Evidence of other etiology than AA for bone marrow failure, including positive clastogenic stress cytogenetic assay for Fanconi anemia and marrow chromosome abnormalities typical of myelodysplasia.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2000-03-17; Primary Completion 2003-12-09 (Actual); Study Completion 2015-05-12 (Actual)

PRIMARY OUTCOMES:
reduction in 24-month relapse | 24 months
  reduction in 24-month relapse

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS. Acquired aplastic anemia. JAMA. 1999 Jul 21;282(3):271-8. doi: 10.1001/jama.282.3.271. No abstract available. PMID 10422997
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Nimer SD, Ireland P, Meshkinpour A, Frane M. An increased HLA DR2 frequency is seen in aplastic anemia patients. Blood. 1994 Aug 1;84(3):923-7. PMID 8043874
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-H-0032.html